CLINICAL TRIAL: NCT02874456
Title: Pilot Study to Detect Zika Virus in Sperm
Acronym: ZIKSPERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Centre Hospitalier Universitaire de la Guadeloupe (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/16/7941
Record Dates: First submitted 2016-05-06; First posted 2016-08-22 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Viruses
Keywords: Zyca virus
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virus detection (Experimental): detection of ZIKA virus in blood and sperm
  Interventions: Other: virus detection

INTERVENTIONS:
Other: virus detection — Men will give semen, urine and blood specimens 7 days after the beginning of clinical signs and 11, 20, 30, 60 and 90 days after. ZIKV RNA will be detected in seminal plasma, native semen cells and processed spermatozoa.

SUMMARY:
The purpose of this study is to seek the presence of ZIKV in semen, to determine its localization and to assess the efficiency of spermatozoa processing methods to obtain virus free spermatozoa.

DETAILED DESCRIPTION:
Since the end of 2015 an epidemic of ZIKA virus (ZIKV) infections is occurring in the Antilles-Guyana departments and focuses our attention on ZIKV and the risk of transmission during assisted reproductive technologies (ART). The importance of this epidemic and the presence in mainland of its mosquito vector (Aedes albopictus) point out the risk of a geographic extension of this infection. In this context the use of Medically Assisted Procreation leads to several questions when patients are infected. The question surges for patients (women and men) who live in epidemic areas but also for people who return from these regions and many other countries within the epidemic area (principally south and central America) and who need ART. Information about localization of ZIKV in the genital tract or shedding is poorly documented. Only two case reports detected ZIKV RNA in the semen and a sexual transmission was described. However, there is no data on the duration of the presence of ZIKV in semen and on localization of ZIKV in semen compartments (cells, seminal plasma, spermatozoa). The purpose of this study is to seek the presence of ZIKV in semen, to determine its localization and to assess the efficiency of spermatozoa processing methods to obtain virus free spermatozoa.

This is a prospective study involving 15 patients, with acute ZIKV infection and a positive RNA detection in blood or/and urines (Institut Pasteur, Pointe-à-Pitre). Men will give semen, urine and blood specimens 7 days after the beginning of clinical signs and 11, 20, 30, 60 and 90 days after. ZIKV RNA being diagnosed with blood and/or urine sample positive for ZIKV RNA. ZIKV RNA will be detected in seminal plasma, native semen cells and processed spermatozoa. Semen sampling and processing will be performed within the ART laboratory of the hospital of Pointe-à-Pitre (Guadeloupe) and research of ZIKV RNA in the laboratory of Virology of Toulouse University Hospital. This study will identify the presence or absence of ZIKV seminal shedding and in case of shedding, verify the efficiency of semen processing to obtain virus free spermatozoa.

These results are important to understand the physiopathology of ZIKV infection and will help to define the management and viral safety procedures during Medically assisted Procreation in the context of ZIKV epidemic.

ELIGIBILITY:
Inclusion Criteria:

* infection by ZIKA virus in early stage

Exclusion Criteria:

* non infected male,
* erection problems

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
presence of Zika virus on RNA by polymerase chain reaction | 6 months
  Presence or absence of ZIKV seminal shedding and in case of shedding, verify the efficiency of semen processing to obtain virus free spermatozoa.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bujan, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Joguet G, Mansuy JM, Matusali G, Hamdi S, Walschaerts M, Pavili L, Guyomard S, Prisant N, Lamarre P, Dejucq-Rainsford N, Pasquier C, Bujan L. Effect of acute Zika virus infection on sperm and virus clearance in body fluids: a prospective observational study. Lancet Infect Dis. 2017 Nov;17(11):1200-1208. doi: 10.1016/S1473-3099(17)30444-9. Epub 2017 Aug 23. PMID 28838639